CLINICAL TRIAL: NCT03904199
Title: A Prospective Randomized Study of a Personalized Approach to the Inpatient Management of Hospitalized Oncology Patients With Hyperglycemia
Brief Title: Prospective Study of Personalized Approach to Inpatient Patients With Hyperglycemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-19637
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Hyperglycemia
Keywords: High Blood Sugar; High Blood Glucose
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Basal-Prandial-Correctional Insulin Regimen (Experimental): Participants hospitalized in the medical, hematologic, or bone marrow transplant units will begin with basal long-acting insulin glargine with correctional and prandial rapid-acting insulin that is personalized and precise, to achieve target blood glucose levels with daily assessments during hospitalization. Adjustments will be made in real time to reach the target range.
  Interventions: Drug: Insulin
- Standard of Care Insulin Regimen (Active Comparator): Participants hospitalized in the medical, hematologic, or bone marrow transplant units' blood sugar levels will be managed with sliding scale insulin or a combination of long- and short-acting insulin as per standard of care.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Participants will receive long-acting insulin and/or rapid-acting insulin per protocol
  Other Names: Basal insulin; Prandial insulin

SUMMARY:
The purpose of this study is to compare the outcomes between hospitalized cancer patients with high blood sugar receiving the current standard of care of administering insulin, and hospitalized cancer patients receiving a new, individualized method of insulin administration.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Provide race and ethnicity information
* Male or female, aged 18 years or greater
* Diagnosed with cancer
* Hospitalized at MCC in the medical, hematologic, or bone marrow transplant units
* Having in-hospital hyperglycemia with or without a pre-existing diagnosis of DM, with 2 measurements of BG > 180 mg/dL and/or 1 measurement of BG > 350mg/dL within the first 72 hours of admission, detected by bedside point-of-care testing and/or basic metabolic panel laboratory data.
* Participants enrolled in other clinical trials are admissible to this trial.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:
* Participants < 18 years of age
* Participants at the end of life and/or with limited life expectancies (< 6 months)
* Participants without cancer diagnoses
* Surgical patients and patients admitted directly to the intensive care unit, other than those in the Bone Marrow Transplant Unit, who are included
* Participants treated and discharged in outpatient settings (ie, direct referral center, infusion center, or clinical research unit) or those admitted for observation only (hospitalized less than 24 hours)
* Participants on total parenteral nutrition
* Participants on insulin pumps
* Participants admitted with diabetic ketoacidosis and hyperglycemic hyperosmolar syndrome
* Pregnant Participants based on medical history
* Participants being followed by endocrinology for hyperglycemia or hypoglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Proportion of blood glucose values within normal range | During hospital admission, up to 30 days
  Proportion of blood glucose values in the 70 mg/dL to 180 mg/dL (normal) range

SECONDARY OUTCOMES:
Proportion of high blood glucose levels | During hospital admission, up to 30 days
  Proportion of blood glucose values >180 mg/dL
Proportion of low blood glucose levels | During hospital admission, up to 30 days
  Proportion of blood glucose values <70 mg/dL
Duration of normal blood glucose level | During hospital admission, up to 30 days
  Duration of blood glucose values in the 70 mg/dL to 180 mg/dL (normal) range

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Pabbathi, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No